CLINICAL TRIAL: NCT06565455
Title: Growing Healthy Children and Families in Rural Arkansas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 297627
Record Dates: First submitted 2024-08-14; First posted 2024-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Obesity; Health Behavior, Risky
Keywords: Healthy Diet; Community Health; Faith Based Organizations; Cultural Adaptation
MeSH Terms: conditions — Pediatric Obesity; Health Risk Behaviors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Seven healthy eating modules, delivered by Community Health Workers (CHW) in the home setting, for 14 weeks. Plus two to three cooking demonstration in the church setting.
  Interventions: Behavioral: Growing Healthy Children and Families in Rural Arkansas
- Control/Attention Group (No Intervention): Five video recordings via Facebook/WhatsApp for three months. Video topics:
  * Mental Health
  * Cord Blood Banking
  * Dental Care
  * Immunizations
  * Behavioral Problems in Children

INTERVENTIONS:
Behavioral: Growing Healthy Children and Families in Rural Arkansas — The intervention will consist of seven healthy eating culturally developed modules, which will be implemented/delivered in the participants home and two cooking demonstration/tasting workshops for the participants in the intervention group (mothers in the church setting and individual and collective goal settings for the intervention group.
  Arms: Intervention Group

SUMMARY:
Childhood obesity is a national problem with racial and ethnic disparities specifically among Hispanic children. The primary purpose of this study is to develop and implement a culturally appropriate healthy eating intervention called Growing Healthy Children and Families in Rural Arkansas.

Specific Aim (SA) 1. To develop a culturally appropriate healthy eating promotion intervention (Growing Healthy Children and Families in Rural Arkansas) in collaboration with Hispanic churches and their congregants.

SA2. To conduct the Growing Healthy Children and Families in Rural Arkansas intervention in eight churches (four churches in the intervention vs four in the control/attention group), and to assess the feasibility and acceptability of implementing the intervention.

SA3. To assess the impact of the Growing Healthy Children and Families in Rural Arkansas intervention on healthy food preparation (mothers) and intake of fruits and vegetables (child).

The investigators will compare between the intervention group (16 mother-child dyads) versus the control/attention group (16 mother-child dyad) to see if the intervention is effective in improving diet quality and changing cooking behaviors.

Participants will:

1. Participate in cooking workshops and one to one learning activities
2. Report on diet and physical activity
3. Will measure fruit and vegetable intake

DETAILED DESCRIPTION:
The primary purpose of this study is to develop and implement a culturally appropriate healthy eating intervention called Growing Healthy Children and Families in Rural Arkansas , to be delivered in the home and church setting by lay Community Health workers (CHW).

Specific Aim (SA) 1. To develop a culturally appropriate healthy eating promotion intervention (Growing Healthy Children and Families in Rural Arkansas ) in collaboration with Hispanic churches and their congregants (formative).

SA2. To conduct the Growing Healthy Children and Families in Rural Arkansas intervention in eight churches (four churches in the intervention vs four in the control/attention group), and to assess the feasibility and acceptability of implementing the intervention (implementation).

SA3. To assess the impact of the Growing Healthy Children and Families in Rural Arkansas intervention on healthy food preparation (mothers) and intake of fruits and vegetables (child).

To achieve Aim 1, Healthy eating culturally adapted modules will be developed from existing sources The healthy eating modules will consist of: Cause and long-term consequences of childhood obesity, Importance of hydration , Physical Activity, Recommended meal portions and meal planning, Sugar Smart, Ultra-processed foods, Fruits and vegetables.

The investigators will recruit up to 15 women to participate in focus groups (FGs) to participate in an iterative process of culturally adapting the healthy eating modules. FGs will be audio-recorded on Zoom or on an encrypted iPad, and professionally transcribed for data analysis. A moderator will lead the FGs, and a note taker will be present during the FGs.

To achieve aim 2, the investigators will recruit and train 10 lay CHWs to deliver the intervention. Priest, pastors, sisters, and/or church staff will approach women who are active in the church setting to discuss the program goals and assess their interest in becoming CHWs. The training will consist of learning the 7 learning modules, and how to effect and motivate behavior change.

Hispanic mother and-child dyads will be recruited to participate in the Growing Healthy Children and Families in Rural Arkansas intervention via word or mouth from priests, sisters, and church staff and via fliers being posted in the churches. The objective is to recruit a total of 16 mother-child dyad, for the intervention group and 16 mother-child dyads for the control/attention group. The total sample, size will be 64 participants.

Randomization will occur at the level of the church. Each dyad will be assigned to either the Growing Healthy Children and Families in Rural Arkansas intervention group or the control group. The Growing Healthy Children and Families in Rural Arkansas intervention group will be implemented at home by the lay CHW bi-weekly for 14 weeks. Participants within the Growing Healthy Children and Families in Rural Arkansas intervention will also attend two Cooking Demonstrations/Tasting Workshops. The workshops will be led by the CHW Specialist, and the dietitian. The workshops are projected to last 2-3 hrs. 60 minutes for teaching nutrition facts, healthy ingredient selection, portion sizes, and the nutritional value of typical Hispanic dishes. The remaining 60-90 minutes will be dedicated to cooking.

The control group will receive seven bi-weekly messaging videos for 12 weeks via Facebook/whatsApp. The messaging videos will last 5-15 minutes and will be delivered in Spanish or English. The topics of the messaging videos are as follows: Mental health issues that affect the Hispanic community, childhood vaccinations Cord blood banking, recommended adult vaccinations, common childhood diseases, dental care for adults and children common behavioral problems in children.

To achieve Aim 3, the investigators will test differences between the intervention and control groups. To determine if there is a change in food preparation in the home setting by the participant (mother) the investigators will measure home cooking quality at T0, and T1. The instrument to evaluate if there is a difference after implementation of the Growing Healthy Children and Families in Rural Arkansas intervention is the HCQ2. To assess if there is a change in intake of fruits and vegetables, in children that participated in the Growing Healthy Children and Families in Rural Arkansas intervention and the control/attention group the investigators will use the Veggie Meter and the Block FFQ at T0 and T1.

The investigators will use descriptive statistics to describe our sample and to make comparisons between the intervention and control/attention group. For the primary outcomes, of changes in dietary behaviors at the family level and change in diet quality, the investigators will use pre-post data (T0 and TI). Secondary outcomes of consumption of fruits and vegetables, consumption of sugar drinks, and physical activity, will be analyzed by using an analysis of covariance (ANCOVA) model from baseline T0, to T1 in children and mothers in both groups.

Data analysis of the FGs qualitative data: FGs transcripts will be uploaded to MAXQDA software for data management and to analyze the transcripts. The investigators will use Rapid analytical techniques to code and uncover themes in the transcripts.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45 years old
* Living in the United States for at least one year
* At least one child aged 7 to 12 years old, and
* English and/or Spanish speaker

Exclusion Criteria:

* Unable to read or write in English or Spanish.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Mothers should be any women who self identifies as Hispanic from Mexico, Central Puerto Rico, and South America.
  Children can be either gender.
Enrollment: 64 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Changes in dietary behavior | Baseline (T0), Week 22 (T1)
  Evaluated via eating habits as reported through the Food Frequency Questionnaire
Change in diet quality - Food Frequency Questionnaire | Baseline (T0), Week 22 (T1)
  Evaluated based on eating habits reported through the Food Frequency Questionnaire
Change in diet quality - Healthy Cooking Questionnaire-2 | Baseline (T0), Week 22 (T1)
  Evaluated based on eating habits reported through the Healthy Cooking Questionnaire-2

SECONDARY OUTCOMES:
Consumption of fruits and vegetables | Baseline (T0), Week 22 (T1)
  Evaluated through the Veggie Meter measures
Consumption of sugary drinks | Baseline (T0), Week 22 (T1)
  Evaluated through the FFQ
Physical activity | Baseline (T0), Week 22 (T1)
  Evaluated through the PA Screener

CONTACTS AND LOCATIONS:
Overall Officials: Martha Rojo, PhD, Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No